CLINICAL TRIAL: NCT06943313
Title: 68Ga-Labeled pAKTi Molecular Probe Combined With PET/CT for Breast Cancer Imaging
Brief Title: Breast Cancer PET/CT Imaging With 68Ga-pAKTi
Status: Enrolling by invitation | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Shaoli Song, PhD, Professor, Fudan University
Other Study IDs: 2503317-27
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancers; PIK3CA Mutation-Related Tumors; PI3K Pathway Activated Tumors; PET / CT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: 68Ga-pAKTi PET/CT probe — A total of 20 patients with breast cancer will be enrolled. Screening will be conducted within 14 days prior to administration of 68Ga-pAKTi (from Day -14 to Day -1). Subjects who meet all inclusion criteria and none of the exclusion criteria will receive an intravenous injection of 68Ga-pAKTi on Day 0, followed by PET/CT imaging.

SUMMARY:
Abnormal activation of the PI3K-AKT signaling pathway in breast cancer patients is closely associated with tumor progression. Phosphorylated AKT (p-AKT) serves as a key indicator of pathway activation. In this study, we utilize a novel probe, 68Ga-pAKTi, which enables precise targeting of tumor p-AKT expression levels to monitor PI3K-AKT pathway activation. The aim of this study is to evaluate the diagnostic accuracy of 68Ga-pAKTi PET/CT in detecting p-AKT expression in breast cancer and to compare its performance with that of 18F-FDG PET/CT.

A total of 20 patients with breast cancer will be enrolled. Screening will be conducted within 14 days prior to administration of 68Ga-pAKTi (from Day -14 to Day -1). Subjects who meet all inclusion criteria and none of the exclusion criteria will receive an intravenous injection of 68Ga-pAKTi on Day 0, followed by PET/CT imaging. Biopsy/pathological results and conventional imaging findings will be followed up to validate the diagnostic efficacy of 68Ga-pAKTi PET/CT in accurately detecting p-AKT expression in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signs the informed consent form.
2. Age ≥ 18 years.
3. Pathologically confirmed or highly suspected breast cancer based on conventional imaging.
4. Estimated life expectancy > 3 months as determined by the physician.
5. Agrees to practice strict contraception for at least 28 days following the PET/CT examination.
6. Willing and able to comply with the study protocol.
7. Has not undergone surgical resection of the lesion.
8. Has participated in molecular testing at the Precision Oncology Center of Fudan University Shanghai Cancer Center, and harbors a PIK3CA mutation, PTEN mutation, or upregulation of the PI3K-AKT-mTOR pathway.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Unable to lie still on the PET/CT scanner bed during the examination or intolerant to PET imaging.
3. Participation in another interventional clinical trial within 1 month prior to screening.
4. Patients who are lost to follow-up.
5. Any other condition that, in the opinion of the investigator, may interfere with the study or make the subject unsuitable for participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value | From enrollment to the end of imaging at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China